CLINICAL TRIAL: NCT04473924
Title: Standard Therapy or Individualized Immunosuppression For Lowering Adverse Event Risk
Acronym: STIFLE-RISK
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has never started as sponsor did not approve for funding.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-31500
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Infection; Transplant;Failure,Kidney
MeSH Terms: conditions — Infections | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Body surface area-based mycophenolate dosing (Experimental): Intervention group will receive mycophenolate mofetil 750 mg/m^2/day divided into twice daily dosing.
  Interventions: Drug: Mycophenolate Mofetil
- Standard (fixed) dosing (Active Comparator): Active comparator group will receive standard fixed dosing of mycophenolate mofetil 1000 mg twice daily.
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Body surface area-based dosing of mycophenolate
  Other Names: Cellcept
  Arms: Body surface area-based mycophenolate dosing
Drug: Mycophenolate Mofetil — Standard (fixed) dosing of mycophenolate
  Other Names: Cellcept
  Arms: Standard (fixed) dosing

SUMMARY:
Infections are common and associated with poor outcomes as well as high financial costs after kidney transplantation. Identifying and implementing strategies to reduce infections after kidney transplantation is important for improving patient outcomes. This study seeks to determine the feasibility of body surface area-based dosing of mycophenolate compared to standard dosing of mycophenolate in a pilot randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult transplant recipients ≥18 years of age who have a functional allograft and have undergone kidney transplantation between six months and two years prior to study enrollment
* Receiving mycophenolate mofetil for maintenance transplant immunosuppression at the time of the screening visit

Exclusion Criteria:

* Evidence of rejection on routine six month post-transplant biopsy
* Prior intolerance to mycophenolate mofetil necessitating drug discontinuation
* Are or are planning to become pregnant, due to inability to take mycophenolate
* Are marginally housed, due to concerns regarding routine follow-up
* Are actively participating in a different interventional trial that may affect immunosuppression dosing
* Are unwilling to consent to participate
* Institutionalized individuals or prisoners
* Are actively abusing illicit drugs or alcohol
* Have a history of poor or doubtful compliance (e.g., frequently missed appointments)
* Have cognitive impairment prohibiting participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate in a trial of BSA-based vs. fixed dosing of mycophenolate | 6 months
  Assess the ratio of participants screened to enrolled into the study

SECONDARY OUTCOMES:
Feasibility of a trial of BSA-based vs. fixed dosing of mycophenolate | 6 months
  Assess the rate of dropout from the study
Collect pilot data of efficacy in a trial of BSA-based vs. fixed dosing of mycophenolate | 6 months
  Collect pilot data on number of overall hospitalizations
Collect pilot data of efficacy in a trial of BSA-based vs. fixed dosing of mycophenolate | 6 months
  Collect pilot data on infectious-related hospitalizations
Collect pilot data of efficacy in a trial of BSA-based vs. fixed dosing of mycophenolate | 6 months
  Collect pilot data on incidence of leukopenia

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Ku, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No